CLINICAL TRIAL: NCT04764838
Title: The Effect of Yoga on Sexual Function in Primiparous Pregnants: Single-Blind Randomized Controlled Study
Brief Title: The Effect of Yoga on Sexual Function in Primiparous Pregnants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Halic University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: Yoga on Sexual Function
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Pregnancy Related; Sexual Dysfunction; Exercise
Keywords: pregnancy; Sexual function; yoga
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Motor Activity | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Randomized controlled single blind
Who Masked: Investigator, Outcomes Assessor
Masking Description: Will not be shared with other researchers and statisticians related to the intervention and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervantion (Experimental): Pregnant Yoga
  Interventions: Other: Yoga
- Control (No Intervention): The clinic will receive routine care

INTERVENTIONS:
Other: Yoga — Breath Awareness Training (5 minutes) Asanas (20 minutes)
  * Bending sideways in Mountain Stance
  * Standing Pelvic Shaking Warrior Stance II Squatting and malasana (wreath pose) Breath awareness in lotus pose (sitting) Cane pose Fixed Butterfly / Angel Pose
  * Sitting wide in Angel Pose Cat Pose Tiger Breath Mudra and meditation (10 minutes)
  Arms: Intervantion

SUMMARY:
This study was planned as a single blind randomized controlled type in order to examine the effect of yoga on sexual function in primipara pregnant women.150 pregnant women will be randomized.The data will be interviewed online with pregnant women and online yoga training will be held for the intervention group

DETAILED DESCRIPTION:
This study was planned as a single blind randomized controlled type in order to examine the effect of yoga on sexual function in primipara pregnant women. The data of the research will be collected through the "Data Collection Form, Female Sexual Function Scale (FSFI)" and The Body Exposure During Sexual Activities Questionnaire (BESAQ), which are created by the researchers by scanning the literature. Research Volunteers who apply to SBU Haseki Training and Research Hospital Pregnancy Outpatient Clinic and meet the sample selection criteria will constitute the sample of the study. In order to determine the minimum sample size required for this study, the power analysis 80% power and α = 0.50 were calculated to include a total of 138 women with a minimum 69 sample size in each group. The intervention and control ratio is 1. However, considering the probability of loss, 150 pregnant women will be randomized. The data will be interviewed online with pregnant women and online yoga training will be held for the intervention group, and the data will be uploaded to the ISM SPSS 22.0 (Statistical Package for the Social Sciences) statistics program; Parametric (Anova and T test) and nonparametric (Mann-Whitney U Test, Kruskal Wallis, Chi Square) statistical methods will be used.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,

  * In primiparous pregnant women (18-26 weeks),
  * Female Sexual Function Scale (FSFI) score> 22.7,
  * Volunteering to participate in research,
  * To speak Turkish.

Exclusion Criteria:

* Having a disability that makes it difficult for the pregnant woman to do yoga asanas,

  * have done yoga Subtraction criterion Not attending the trainings regularly,
  * Not attending at least 5 of the trainings

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant
Enrollment: 150 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
sexual function | 4 weeks
  FSFI(FEMALE SEXUAL FUNCTION INDEX)

SECONDARY OUTCOMES:
Body ımage | 4 weeks
  BESAQ (The Body Exposure during Sexual Activities Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Şule Tanrıverdi, MsC, Principal Investigator — Haseki Hospital
Locations (1):
- Haseki Hospital, Sultangazı, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This study was planned as a single blind randomized controlled type in order to examine the effect of yoga on sexual function in primipara pregnant women.150 women were randomized. Pregnant women in the intervention group are applied online yoga, and pregnant women in the control group receive clinical routine care.
Supporting Information: Study Protocol
Time Frame: January-June ( 6 monts)